CLINICAL TRIAL: NCT03236428
Title: A Phase II Study of the CD38 Antibody Daratumumab in Patients With High-Risk MGUS and Low-Risk Smoldering Multiple Myeloma
Brief Title: Phase II Study of the CD38 Antibody Daratumumab in Patients With High-Risk MGUS and Low-Risk Smoldering Multiple Myeloma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Janssen Pharmaceuticals (Industry); Multiple Myeloma Research Consortium (Network); Blood Cancer Research Partnership (Other); The Leukemia and Lymphoma Society (Other)
Responsible Party: Principal Investigator, Irene Ghobrial, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-212
Record Dates: First submitted 2017-07-11; First posted 2017-08-01 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Monoclonal Gammopathy; Smoldering Multiple Myeloma
Keywords: Smoldering Multiple Myeloma; Monoclonal Gammopathy
MeSH Terms: conditions — Paraproteinemias; Smoldering Multiple Myeloma | interventions — daratumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Daratumumab (Experimental): Daratumumab will be administered by IV infusion weekly during cycles 1 and 2 Daratumumab will be administered by IV infusion every other week during cycles 3 through 6 Daratumumab will be administered by IV infusion monthly during cycles 7 through 20
  Interventions: Drug: Daratumumab

INTERVENTIONS:
Drug: Daratumumab — Daratumumab is a drug that may kill or stop cancer cells from growing through a variety of mechanisms by attaching to the CD38 molecule
  Other Names: Darzalex

SUMMARY:
This research study is studying a drug as a possible treatment for Monoclonal Gammopathy of Unknown Significance (MGUS) or Smoldering Multiple Myeloma (SMM).

The drug involved in this study is:

-Daratumumab

DETAILED DESCRIPTION:
This research study is a Phase II clinical trial, which tests the effectiveness of an investigational drug. Preliminary experience suggests that daratumumab may prevent or postpone SMM from becoming active multiple myeloma. The purpose of this research study is to determine if the this drug may improve the rate of prevention of multiple myeloma.

Multiple myeloma is a cancer of the plasma cell, which is an important part of the immune system. Patients with active multiple myeloma generally require treatment. There are currently no approved therapies for smoldering multiple myeloma or Monoclonal Gammopathy of Unknown Significance.

Daratumumab is a drug that may kill or stop cancer cells from growing through a variety of mechanisms by attaching to the CD38 molecule, which is over-expressed in multiple myeloma cells. This type of drug is called a monoclonal antibody. The FDA (the U.S. Food and Drug Administration) has not approved Daratumumab for the participant specific disease but it has been approved for use in active Multiple Myeloma.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Must meet criteria for high-risk MGUS or low-risk smoldering myeloma as described below:

High-Risk MGUS

Must have <10% plasma cells and <3.0g/dL M-spike and at least 2 of the following 3 criteria:

* Abnormal free light-chain (FLC) ratio (<0.26 or >1.65)
* M-protein concentration (≥1.5 g/dL)
* Non-IgG M protein (including IgA)

Low-Risk Smoldering Multiple Myeloma

Must only present with 1 of the following criterion:

* Monoclonal Protein ≥ 3 g/dL

  ---≥ 10% Bone Marrow Plasma Cells
* FLC ratio < 0.125 or > 8

  -No evidence of CRAB criteria† or new criteria of active MM which including the following:
  * Increased calcium levels (corrected serum calcium >0.25 mmol/dL above the upper limit of normal or >0.275 mmol/dL)
  * Renal insufficiency (attributable to myeloma)
  * Anemia (Hb 2 g/dL below the lower limit of normal or <10 g/dL)
  * Bone lesions (lytic lesions or generalized osteoporosis with compression fractures)
  * No evidence of the following new criteria for active MM including the following: Bone marrow plasma cells >60%, Serum involved/uninvolved FLC ratio ≥100, and MRI with more than one focal lesion

    * Participants with CRAB criteria that are attributable to conditions other than the disease under study may be eligible
    * ECOG Performance Status (PS) 0, 1, or 2 (Appendix A)
    * The following laboratory values obtained ≤ 21 days prior to registration:
  * ANC ≥ 1000/uL
  * PLT ≥ 50,000/uL
  * Total bilirubin ≤ 2.0 mg/dL (If total is elevated check direct and if normal patient is eligible.)
  * AST ≤ 3 x institutional upper limit of normal (ULN)
  * ALT ≤ 3 x institutional upper limit of normal (ULN)
  * Creatinine ≤ 2 mg/dL or Creatinine Clearance ≥ 40 mL/min

    * Ability to understand and the willingness to sign an informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care.
    * Female patients who are postmenopausal for at least 1 year before the screening visit or are surgically sterile are eligible. Females of childbearing potential (as defined below) may also be eligible but must have a negative serum or urine pregnancy test with a sensitivity of at least 25 mIU/mL within 21 days of registration.
  * A female of childbearing potential is a sexually mature female who:
* Has not undergone a hysterectomy (the surgical removal of the uterus) or bilateral oophorectomy (the surgical removal of both ovaries)

OR

---Has not been naturally postmenopausal (amenorrhea following cancer therapy does not rule out childbearing potential) for at least 24 consecutive months (i.e., has had menses at any time during the preceding 24 consecutive months)

Exclusion Criteria:

* Any prior therapy for symptomatic Multiple Myeloma or smoldering Multiple Myeloma should also be excluded, including prior use of IMIDs, proteasome inhibitors, or CD138 inhibitors. Prior therapy for smoldering Multiple Myeloma with agents that are not therapeutically active against MM is not an exclusion criterion.
* Other concurrent chemotherapy, immunotherapy, radiotherapy, or any ancillary therapy considered investigational. Prior therapy with bisphosphonates is allowed. Prior radiation therapy to a solitary plasmacytoma is allowed.
* Concurrent exposure to any commercially available agents known to be active against SMM and MM.
* Serious medical or psychiatric illness likely to interfere with participation in this clinical study.
* Diagnosed or treated for another malignancy within 2 years of enrollment, with the exception of complete resection of basal cell carcinoma or squamous cell carcinoma of the skin, an in situ malignancy, or low-risk prostate cancer after curative therapy.
* Subject has known chronic obstructive pulmonary disease (COPD) with a Forced Expiratory Volume in 1 second (FEV1) < 50% of predicted normal.
* Note that FEV1 testing is required for patients suspected of having COPD and subjects must be excluded if FEV1 <50% of predicted normal.

  * Subject has known moderate or severe persistent asthma within the past 2 years or currently has uncontrolled asthma of any classification.
  * Subjects who currently have controlled intermittent asthma or controlled mild persistent asthma are allowed in the study
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, uncontrollable cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant or nursing women will be excluded from the study.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to Daratumumab.
* Known seropositive for or active viral infection with human immunodeficiency virus (HIV), hepatitis B virus (HBV) or hepatitis C virus (HCV). Patients who are seropositive because of hepatitis B virus vaccine are eligible. Patients who are positive for hepatitis B core antibody or hepatitis B surface antigen must have a negative polymerase chain reaction (PCR) result before enrollment. Those who are PCR positive will be excluded.
* Major surgery within 4 weeks before enrollment.
* Subject is known or suspected of not being able to comply with the study protocol (eg, because of alcoholism, drug dependency, or psychological disorder). Subject has any condition for which, in the opinion of the investigator, participation would not be in the best interest of the subject (eg, compromise the well-being) or that could prevent, limit, or confound the protocol-specified assessments.
* Vaccination with live attenuated vaccines within 4 weeks of first study agent administration
* Subject has clinically significant cardiac disease, including significant ischemic coronary disease, congestive heart failure (New York Heart Association [NYHA] Class III or IV), unstable arrhythmias, myocardial infarction or unstable angina within 6 months before randomization, a history of additional risk factors for torsades de pointes (eg, electrolyte abnormalities, family history of Long QT Syndrome), or a family history of sudden cardiac death before age 40.
* Participation in other therapeutic clinical trials, including those with other investigational agents not included in this trial, within 30 days of the start of this trial and throughout the duration of this trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2017-11-24 (Actual); Primary Completion 2026-10-04 (Estimated); Study Completion 2026-10-04 (Estimated)

PRIMARY OUTCOMES:
The Proportion Of Patients In Deep Response | 2 years
  To determine the proportion of patients who are in VGPR or better after twenty cycles of therapy with Daratumumab. This will be determined at the time of best overall response. The estimate and the two-sided 90% binomial confidence interval will be provided in the analysis.

SECONDARY OUTCOMES:
Objective Response Rate | 2 years
  The objective response rate (partial response or better according to the modified IMWG criteria) and the proportion of patients with a MRD, CR, PR or MR will be reported with 90% exact binominal confidence interval (CI). The exact two-sided 90% CI around response rate will be no wider than 28% with 40 eligible patients.
Duration of Response | 2 years
  To estimate the duration of response (time from objective response to disease progression or death, or date last known progression-free and alive for those who have not progressed or died) the Kaplan-Meier method will be used.
Complete Response Rate | 2 years
  The duration of overall CR is progression or death. Patients who have not progressed or died are censored at the date last known progression-free.
Overall Response Rate | 2 years
  The duration of overall response is measured as the time from initiation of first response to first documentation of disease progression or death. Patients who have not progressed or died are censored at the date last known progression-free.
Progression Free Survival | 2 years
  PFS is defined as the time from first-dose to the disease progression or death from any cause. Patients who have not progressed or died are censored at the date last known progression-free.
Incidence of Treatment Emergent Adverse Events (Safety and Tolerability) | 2 years
  Safety analysis will be conducted using the Safety Population defined as any patient receiving one dose of study treatment. For toxicity reporting, all adverse events and laboratory abnormalities will be graded and analyzed using CTCAE version 4 as appropriate.

CONTACTS AND LOCATIONS:
Overall Officials: Irene Ghobrial, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (6):
- United States (6):
  - Pacific Cancer Care, Monterey, California
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Karmanos Cancer Insitute, Detroit, Michigan

IPD SHARING:
Plan to Share IPD: No